CLINICAL TRIAL: NCT07260929
Title: VR Goggles-Supported Virtual Reality Model in Midwifery Basic Clinical Skills Training: A Randomized Controlled Trial
Brief Title: VR Goggles-Supported Virtual Reality Model in Midwifery Basic Clinical Skills Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ezgi Dirgar, Associate Professor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/317
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Clinical Skills Training; Midwifery Education
Keywords: Midwifery education; clinical skills training; virtual reality-based learning; simulation-based training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (VR Goggle-Assisted VR Training) (Experimental): Participants in this arm will receive basic clinical skills training using a VR goggle-supported virtual reality model specifically designed for midwifery education. The VR module includes interactive simulations, step-by-step procedural guidance, and scenario-based skill practice. Training will be delivered individually under supervision and will cover essential midwifery clinical skills.
  Interventions: Behavioral: VR Goggle-Assisted Simulation Training
- Active Comparator: Traditional Training (Active Comparator): Participants in this arm will receive traditional basic clinical skills training using standard educational methods such as demonstration, skills laboratory practice, and return demonstration. This training follows the current curriculum used in midwifery clinical skills education and does not include virtual reality components.
  Interventions: Behavioral: Standard Clinical Skills Training

INTERVENTIONS:
Behavioral: VR Goggle-Assisted Simulation Training — The VR-based training intervention includes an immersive Virtual Reality clinical skills module delivered through VR goggles. Participants receive structured, scenario-based training covering basic midwifery clinical skills, such as hand hygiene, aseptic technique, vital signs assessment, perineal care, and safe birth positioning. Each session is conducted using interactive 3D simulations that allow learners to observe, practice, and repeat psychomotor and decision-making steps in a risk-free virtual environment. The training is standardized across participants, lasts approximately 30 minutes per session, and is delivered by an instructor trained in VR-assisted education.
  Arms: Experimental (VR Goggle-Assisted VR Training)
Behavioral: Standard Clinical Skills Training — Participants in this Arm will receive standard midwifery basic clinical skills training through conventional laboratory practice without VR exposure. Training content follows the curriculum guidelines and emphasizes hands-on skill development using standard educational materials and instructor demonstrations.
  Arms: Active Comparator: Traditional Training

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of a virtual reality (VR)-based training model supported by VR goggles in improving basic clinical skills among midwifery students. Traditional skills training in midwifery education can be limited by time, instructor availability, and opportunities for repeated practice. VR technology offers an immersive, standardized, and repeatable learning environment that may enhance skill development and learner engagement.

In this study, midwifery students will be randomly assigned to either the VR training group or the traditional training group. Participants in the VR group will practice selected basic clinical skills using a VR goggle-supported simulation model, while the control group will receive standard skills laboratory training. Both groups will be evaluated through objective structured clinical examinations (OSCEs), self-confidence scales, and skill performance checklists.

The study aims to determine whether VR-enhanced training improves clinical skill acquisition, performance accuracy, and learner confidence compared with traditional methods. Findings from this research may help inform modern, technology-supported approaches to midwifery education.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled as an undergraduate midwifery student at Gaziantep University.
* Registered in or scheduled to take the "Basic Clinical Skills" course during the study period.
* Aged 18 years or older.
* Able to provide informed consent and willing to participate throughout the study.
* Has no previous formal training with virtual reality (VR) simulation related to midwifery clinical skills.
* Able to use VR goggles safely (no known conditions that prevent VR use, such as severe motion sickness).

Exclusion Criteria:

* A diagnosed visual, neurological, or vestibular disorder that may interfere with VR use (e.g., epilepsy, severe vertigo).
* A history of severe motion sickness symptoms triggered by digital screens or VR environments.
* Participated previously in a pilot version of the VR training module.
* Currently taking a leave of absence or not actively attending coursework.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Basic Midwifery Clinical Skills Performance | Baseline (pre-training) and immediately post-training (within 1 week after completion of the training program)
  Performance in core midwifery clinical skills (e.g., abdominal examination, Leopold maneuvers, vital signs assessment, hand hygiene, perineal care, and communication skills) will be evaluated using a validated Objective Structured Clinical Examination (OSCE) checklist. Higher scores indicate better skill performance. Student satisfaction and self-confidence in learning will be evaluated using the "Student Satisfaction and Self-Confidence in Learning Scale," which consists of 13 items rated on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 13 (minimum) to 65 (maximum), and higher scores indicate greater satisfaction with the instructional experience and higher self-confidence in learning.

IPD SHARING:
Plan to Share IPD: No